CLINICAL TRIAL: NCT06450431
Title: French Validation of a Specific Tool for Quality of Life Evaluation in Primary Hyperparathyroidism
Brief Title: Parathyroid Assessment of Symptoms French Version
Acronym: PAS_fr
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0151; 2024-A00618-39 (Other: ANSM (IDRCB))
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Quality of Life in Primary Hyperparathyroidism
Keywords: Primary hyperparathyroidism; Parathyroidectomy; Quality of life
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control group: Patients attempting surgical consultation for thyroid nodule, with no history of PHPT.
  Interventions: Other: SF-36 questionnaire French version and PAS.fr questionnaire
- PHPT before surgery group: Patients attempting surgical consultation for PHPT.
  Interventions: Other: SF-36 questionnaire French version and PAS.fr questionnaire
- PHPT 6 months after surgery group: Patients operated for PHPT interrogated 6 months after surgery
  Interventions: Other: SF-36 questionnaire French version and PAS.fr questionnaire
- PHPT 12 months after surgery group: Patients operated for PHPT interrogated 12 months after surgery
  Interventions: Other: SF-36 questionnaire French version and PAS.fr questionnaire
- PHPT 36 months after surgery group: Patients operated for PHPT interrogated 36 months after surgery
  Interventions: Other: SF-36 questionnaire French version and PAS.fr questionnaire

INTERVENTIONS:
Other: SF-36 questionnaire French version and PAS.fr questionnaire — Patients will receive both the SF-36 questionnaire (control generic questionnaire for QoL evaluation validated in French language) and the PAS.fr questionnaire at the designated time (before surgery, 6, 12 or 36 months after surgery) during the consultation, or by mail. For concurrent validation of the PAS.fr questionnaire, a second questionnaire will be sent to the patients 2-4 weeks thereafter.

SUMMARY:
Primary hyperparathyroidism has been associated with an impaired quality of life. Surgery has been suggested to improve this outcome in patients with baseline quality of life impairment; however, few studies have used specific tool for quality of life assessment this pathology, none being validated in French version. The aim of this study is to validate the parathyroid assessment of symptoms (PAS) questionnaire in French language to evaluate quality of life impairment and the impact of surgery in patients with primary hyperparathyroidism.

DETAILED DESCRIPTION:
Besides classic target organs of primary hyperparathyroidism (PHPT) that are the bone and kidneys, patients also present with non-specific and neurocognitive symptoms that impair quality of life (QoL). Several studies have assessed QoL in these patients and the impact of surgery, but using varied tools for QoL evaluation. While observational studies strongly suggest symptoms and QoL improvement after surgery, randomized studies with fewer included patients showed milder results. Therefore, international guidelines have not accepted QoL impairment as an indication for surgery. The reasons of these discrepancies between studies include the use of varied tools to evaluate QoL, either specific or not for this pathology. Using a specific tool for PHPT-related QoL could be more appropriate to understand the impact of surgery; however, no such questionnaire has been validated in French version up today. A specific questionnaire named the parathyroid assessment of symptoms (PAS) has been proposed by the team of J.Pasieka several years ago and has been demonstrated to specifically describe QoL impairment in PHPT based on 13 frequent non-specific symptoms. For the present study, a French version of the PAS (PAS.fr) have been created by double translation followed by a backtranslation that has been validated by the author of the original questionnaire. The aim of this study is to validate the use of PAS.fr in a French population of patients with PHPT to evaluate their QoL impairment and the impact of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PHPT

   * Adult patients
   * Patients with PHPT, whether operated on or not, defined by a calcium level > 2.60 mmol/L with inappropriate PTH (> 15 pg/mL) or normal calcium with elevated PTH (> 65 pg/mL) before surgery.
   * Consulting for PHPT surgery, or at 6, 12, or 36 months post-surgery.
   * Not opposed to participating in the study (questionnaires will be provided/sent with the study information sheet. If the patient returns the questionnaires, it will be considered that they are not opposed to participating in the study).
2. Control Patients

   * Adult patients
   * Patients consulting for thyroid surgery for benign thyroid nodules with normal thyroid function (serum TSH between 0.4 and 4.0 mIU/L) and no hypercalcemia (calcium ≤ 2.6 mmol/L).
   * Not opposed to participating in the study (questionnaires will be provided/sent with the study information sheet. If the patient returns the questionnaires, it will be considered that they are not opposed to participating in the study).

Exclusion Criteria:

* Pregnant women at the time of completing the questionnaires (the child's parathyroid glands can influence the mother's parathyroid status).
* Minors or protected patients (under guardianship/curatorship).
* Patients with secondary/tertiary hyperparathyroidism (defined by hypocalcemia < 2.0 mmol/L with elevated PTH, or hypercalcemia with elevated PTH with a history of kidney transplantation, respectively).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was all patients consulting for PHPT in the surgery department at Nantes University Hospital during the study period:
  In order to study the discriminant validity and specificity of the PAS.fr for PHPT, a control group consisting of euthyroid patients undergoing thyroidectomy for thyroid nodules will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Validate the unidimensionality of the PAS.fr for assessing quality of life in PHPT patients | 4 weeks
  The unidimensionality of the 13 items of the PAS.fr questionnaire will be determined based on their suitability for a confirmatory factor analysis (CFA). Suitability will be judged based on the suitability coefficients RMSEA, TLI and CFI. The adequation will be judged acceptable if RMSEA<0.08, CFI>0.9 and TLI>0.9 and will be judged good if RMSEA<0.05, CFI>0.95 and TLI>0.95.

SECONDARY OUTCOMES:
Reliability of the PAS.fr score | 4 weeks
  Reliability measured by Cronbach's alpha coefficient and McDonald's Omega coefficient. Reliability will be considered acceptable if these coefficients are greater than 0.7 and good if they are greater than 0.8.
Content validity to demonstrate the relevance of the French translation compared to the original version of the PAS.fr | 4 weeks
  Content validity: qualitative validation by the author of the original PAS questionnaire after back-translation of the PAS.fr questionnaire.
Discriminant validity to show that the PAS.fr score is significantly correlated with biological values impacted by PHPT and specific to PHPT | 4 weeks
  Discriminant validation: Spearman correlation between the PAS.fr score and measurements of PTH, calcium, and urinary calcium. Moderate to strong correlations (>0.4) are expected between these values.
Discriminant validity by comparing PAS.fr scores to those of a control population of patients who do not have PHPT | 4 weeks
  Discriminant validation: ANOVA to show differences in PAS.fr scores between HPT1 patients and other patients (control group consisting of patients consulting for thyroidectomy for thyroid nodule (euthyroid)).
Discriminant validity to show that the PAS.fr score can distinguish HPT1 patients with different clinical manifestations | 4 weeks
  Discriminant validation: ANOVA to show differences in the mean PAS.fr scores between a group of HPT1 patients with clinical manifestations (bone involvement defined by the presence of fractures and/or a T-score < -2.5 on bone densitometry and renal involvement defined by the presence of kidney stones < 10 years and/or a glomerular filtration rate < 60 mL/min) and other patients.
Concurrent validation with the SF-36 questionnaire - Reproducibility in stable patients over a period of 15 days | 4 weeks
  Concurrent validation: Spearman correlation coefficients between the PAS.fr score and SF-36 quality of life scores. Weak to moderate positive correlations (>0.2) are expected. - Reproducibility: Intraclass correlation coefficients between PAS.fr scores obtained from two closely timed administrations of the questionnaire (2-3 weeks apart).

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided